CLINICAL TRIAL: NCT06593015
Title: Study Protocol to Redefine Muscle Attenuation Cut-offs for Better Prediction of Mortality in Patients with Cirrhosis: a Comprehensive Post-hoc Validation Study
Brief Title: Protocol for Muscle Attenuation Cut-offs in Cirrhosis
Acronym: Myocirrhosis
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Simone Di Cola, Medical Doctor, University of Roma La Sapienza
Other Study IDs: Prot n 94/19
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cirrhosis; Myosteatosis; Sarcopenia; Sarcopenia in Liver Cirrhosis; Portal Hypertension Related to Cirrhosis; Malnutrition
Keywords: cirrhosis; myosteatosis; cut-offs; diagnosis; sex; muscle attenuation; malnutrition
MeSH Terms: conditions — Fibrosis; Sarcopenia; Malnutrition; Disease; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective cohort: Department of Translational and Precision Medicine, Sapienza University of Rome: The prospective cohort in this study consists of patients with cirrhosis who were prospectively enrolled from 26 different centres across Italy (EpatoSarco groups) between January 2019 and January 2020. The cohort includes a total of 447 patients aged between 40 and 75 years, who underwent abdominal CT scans for various clinical indications. The results of the original study were already published in May 2024.
  Interventions: Diagnostic Test: Radiological tool for the diagnosis of myosteatosis
- Retrospective group: University of Alberta, Edmonton, Alberta, Canada: The retrospective cohort in this study comprises patients with cirrhosis who were evaluated for liver transplantation (LT) at the University of Alberta Hospital in Canada. This cohort includes 1,104 patients who underwent CT imaging as part of their LT evaluation between January 2000 and August 2021. After applying specific exclusion criteria, 863 patients were ultimately included in the analysis. The results of the original study were already published in Apr 2022
  Interventions: Diagnostic Test: Radiological tool for the diagnosis of myosteatosis

INTERVENTIONS:
Diagnostic Test: Radiological tool for the diagnosis of myosteatosis — Calculation of muscle attenuation at L3 CT scan for each patients and evaluation of the relationship between muscle attenuation values and survival
  Groups: Retrospective group: University of Alberta, Edmonton, Alberta, Canada
Diagnostic Test: Radiological tool for the diagnosis of myosteatosis — Calculation of muscle attenuation at L3/L4 CT scan for each patients and evaluation of the relationship between muscle attenuation values and survival
  Groups: Prospective cohort: Department of Translational and Precision Medicine, Sapienza University of Rome

SUMMARY:
The goal of this observational study is to learn if new muscle attenuation cut-offs for the definition of myosteatosis can better predict survival in patients with cirrhosis. The main questions it aims to answer are:

* Can these new muscle attenuation cut-offs more accurately diagnose myosteatosis (fat infiltration in muscle mass ) in cirrhosis?
* Do these cut-offs work effectively across different patient groups, including men and women, those with obesity, and those with fluid retention in the abdomen?

Researchers will compare patients with cirrhosis from a retrospective Canadian cohort to those from a prospective Italian cohort to see if the new cut-offs predict survival better than existing ones**.

Due to the retrospective nature of the study, no action is required from participants.

DETAILED DESCRIPTION:
Detailed Description This observational study seeks to redefine muscle attenuation cut-offs to better predict mortality in patients with cirrhosis, particularly focusing on myosteatosis-a condition characterized by the pathological accumulation of fat within skeletal muscles. Myosteatosis is a critical factor in cirrhosis, associated with poor outcomes, including increased risk of overt hepatic encephalopathy, prolonged hospitalization, post-transplant complications, and reduced survival. The current cut-offs for diagnosing myosteatosis are derived from studies in oncology populations, which may not be appropriate for cirrhosis patients due to specific complications like fluid retention (ascites) and differences in fat and muscle distribution between genders.

Background and Rationale Cirrhosis patients often experience muscle changes due to chronic inflammation and metabolic disturbances, leading to muscle fat infiltration or myosteatosis. This study builds on previous research by Ebadi et al., who proposed sex-specific cut-offs (<33 HU for men and <28 HU for women) for diagnosing myosteatosis based on muscle attenuation values measured via CT scans. However, these cut-offs were derived from a retrospective cohort and have not been validated externally. There is a clear need for liver-specific cut-offs that account for the unique characteristics of cirrhosis, including the impact of fluid retention on BMI and muscle attenuation measurements.

Study Objectives

The primary objective is to validate new muscle mass attenuation cut-offs for the diagnosis of myosteatosis using L3 CT scan evaluations to predict survival and outcomes in patients with cirrhosis. Secondary objectives include:

* Assessing the accuracy of these cut-offs across different patient groups (e.g., by gender, obesity status, and presence of ascites).
* Evaluating the prognostic significance of redefined myosteatosis when combined with sarcopenia (muscle wasting).

Study Design

The study involves a post-hoc analysis of data from two large cohorts:

1. Retrospective Cohort (Canada): This cohort consists of 1,104 patients evaluated for liver transplantation (LT) at the University of Alberta Hospital between January 2000 and August 2021. After applying exclusion criteria (e.g., absence of cirrhosis, multi-organ transplantation), 863 patients were included in the final analysis.
2. Prospective Cohort (Italy): This cohort includes 447 patients from 26 Italian centers, prospectively enrolled between January 2019 and January 2020, with cirrhosis who underwent abdominal CT scans. After excluding patients with incomplete data, 433 patients were included in the analysis.

Data Collection

Data were collected at the time of enrollment and included:

* Demographic characteristics: Age, sex
* Anthropometric measurements: Height, weight, BMI
* Cirrhosis etiology: Hepatitis C, alcohol-related liver disease, non-alcoholic steatohepatitis (NASH), etc.
* Comorbidities: Diabetes, hypertension, dyslipidemia
* Liver complications: Refractory ascites, variceal bleeding, hepatic encephalopathy, hepatocellular carcinoma (HCC)
* Liver classification and blood tests: Child-Pugh score, MELD score, MELD-Na score, albumin, sodium, creatinine, INR, bilirubin, hemoglobin, etc.
* Radiological evaluation: Muscle mass and quality assessments via CT scans at the L3 or L3/L4 vertebrae level, including muscle attenuation and skeletal muscle index (SMI).

Radiological Assessment Muscle mass and attenuation were measured using CT scans, with radiodensity (measured in Hounsfield Units, HU) being the primary indicator of myosteatosis. The HU thresholds for assessing skeletal muscle ranged from -29 to +150 HU. The muscle area was adjusted for height to obtain the L3 or L3/L4 skeletal muscle index (SMI). Sarcopenia was diagnosed using validated SMI cut-off values (<50 cm²/m² for men and <39 cm²/m² for women). The study specifically examines muscle attenuation in relation to BMI, gender, and ascites to refine the diagnostic criteria for myosteatosis.

Patient Classification

Patients were classified into four groups based on the presence of myosteatosis and sarcopenia:

1. No muscle changes: No myosteatosis, no sarcopenia.
2. Isolated myosteatosis: Myosteatosis without sarcopenia.
3. Isolated sarcopenia: Sarcopenia without myosteatosis.
4. Combined: Both myosteatosis and sarcopenia.

Statistical Analysis

To validate the new cut-offs, the study will:

* Perform univariate analyses on variables likely associated with mortality, such as muscle attenuation and muscle mass.
* Conduct multivariate analyses to assess the impact of confounding variables.
* Use Receiver Operating Characteristic (ROC) curves, stratified by sex, BMI, and ascites, to identify the muscle attenuation values most strongly associated with mortality.
* Assess non-causal concordance (kappa index) between CT scan measurements across the two cohorts by exchanging and reanalyzing a subset of data.

The study aims to confirm or refine the cut-offs proposed by Ebadi et al. and evaluate their adequacy in different cirrhotic populations, stratified by disease severity and history of decompensation.

Follow-Up and Outcomes In the retrospective cohort, patients were followed for an average of 24 ± 35 months, with outcomes such as death and liver transplantation recorded. In the prospective cohort, patients were followed for 12 months post-enrollment, with outcomes including survival, hospitalizations, and liver-related complications. Data from these follow-ups will be crucial in validating the predictive power of the new muscle attenuation cut-offs.

Ethical Considerations

The study protocol has been reviewed and approved by the Institutional Review Board of the University of Alberta (approval number: Pro00066572) for the retrospective cohort and by the Ethical Committee of the Rome's Center (EC n° 94/19 30/01/19) for the prospective cohort. Each participating center provided its own ethical approval, and all patients gave informed consent for their participation.

Conclusion This study aims to provide a more accurate and tailored method for diagnosing myosteatosis in patients with cirrhosis by refining muscle attenuation cut-offs. By validating these new thresholds, the study hopes to improve the prediction of patient outcomes and aid in the management and treatment strategies for cirrhosis, ultimately leading to better patient care and survival rates.

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort:

* Clinical, radiological and/or histological diagnosis of cirrhosis
* Abdominal CT-scan obtained as part of the LT evaluation

Prospective cohort:

* Clinical, radiological and/or histological diagnosis of cirrhosis
* Age 40-75 years
* Abdominal CT-scan

Exclusion Criteria:

Retrospective cohort:

* Multi-organ transplantation
* Re-transplantation

Prospective cohort:

* Patient on LT waiting lists
* Hepatocellular carcinoma (HCC)
* History of LT
* Concomitant neuromuscular disease
* Current malignancy other than non-melanocytic skin cancer
* History of serious extrahepatic disease
* HIV infection.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective cohort, 1104 patients were evaluated for LT between January 2000 and August 2021 in the University of Alberta Hospital (Canada), of whom 241 were excluded for not meeting the inclusion and exclusion criteria, so 863 patients were considered for the analysis.
  In the prospective cohort, 447 patients were prospectively enrolled from 26 Italian centres, 14 of whom were excluded due to incomplete data, leaving 433 patients for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Definition of new L3/L3-L4 muscle attenuation cut-offs to define myosteatosis in relation to risk of death in patients with cirrhosis | 12 months
  The primary outcome is the validation of L3 / L3-L4 muscle attenuation values associated with the overall risk of death. Liver transplantation will be considered as a competing event in any analysis of the clinical impact of muscle damage, according to the above definition and classification.

SECONDARY OUTCOMES:
Association of newly defined myosteatosis with risk of clinical events in patients with cirrhosis | 12 months
  Secondary outcomes: to explore the association between newly defined myosteatosis with the risk of hospitalization for liver related reasons and further decompensation. Hospitalization for liver related reasons will be defined as any hospitalization for any complication of cirrhosis, including day hospital admissions for paracentesis, endoscopic treatments for esophageal varices, trans-jugular intrahepatic porto-systemic shunt.
  Further decompensation will be defined according to the BavenoVII criteria (ref)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Translational and Precision Medicine, Sapienza University of Rome, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Given the nature of the databases and the sharing of the project with another centre, we do not believe that individual data can be shared. If necessary, if requested by any author, we can agree on individual data sharing

REFERENCES:
- [Background] Ebadi M, Tsien C, Bhanji RA, Dunichand-Hoedl AR, Rider E, Motamedrad M, Mazurak VC, Baracos V, Montano-Loza AJ. Skeletal Muscle Pathological Fat Infiltration (Myosteatosis) Is Associated with Higher Mortality in Patients with Cirrhosis. Cells. 2022 Apr 14;11(8):1345. doi: 10.3390/cells11081345. PMID 35456024
- [Background] Mehta G, Riva A, Ballester MP, Uson E, Pujadas M, Carvalho-Gomes A, Sahuco I, Bono A, D'Amico F, Vigano R, Diago E, Lanseros BT, Inglese E, Vazquez DM, Sharma R, Tsou HLP, Harris N, Broekhoven A, Kikkert M, Morales SPT, Myeni SK, Riveiro-Barciela M, Palom A, Zeni N, Brocca A, Cussigh A, Cmet S, Escudero-Garcia D, Stocco M, Natola LA, Ieluzzi D, Paon V, Sangiovanni A, Farina E, di Benedetto C, Sanchez-Torrijos Y, Lucena-Varela A, Roman E, Sanchez E, Sanchez-Aldehuelo R, Lopez-Cardona J, Canas-Perez I, Eastgate C, Jeyanesan D, Morocho AE, Di Cola S, Lapenna L, Zaccherini G, Bongiovanni D, Zanaga P, Sayaf K, Hossain S, Crespo J, Robles-Diaz M, Madejon A, Degroote H, Fernandez J, Korenjak M, Verhelst X, Garcia-Samaniego J, Andrade RJ, Iruzubieta P, Wright G, Caraceni P, Merli M, Patel VC, Gander A, Albillos A, Soriano G, Donato MF, Sacerdoti D, Toniutto P, Buti M, Duvoux C, Grossi PA, Berg T, Polak WG, Puoti M, Bosch-Comas A, Belli L, Burra P, Russo FP, Coenraad M, Calleja JL, Perricone G, Berenguer M, Claria J, Moreau R, Arroyo V, Angeli P, Sanchez C, Ampuero J, Piano S, Chokshi S, Jalan R; COBALT Consortium. Serological response and breakthrough infection after COVID-19 vaccination in patients with cirrhosis and post-liver transplant. Hepatol Commun. 2023 Oct 18;7(11):e0273. doi: 10.1097/HC9.0000000000000273. eCollection 2023 Nov 1. PMID 37870985
- [Derived] Di Cola S, D'Amico G, Motamedrad M, Montano-Loza A, Merli M. Study protocol to redefine muscle attenuation cut-offs for better prediction of mortality in patients with cirrhosis: a comprehensive post hoc validation study - a study protocol. BMJ Open. 2025 Mar 25;15(3):e094252. doi: 10.1136/bmjopen-2024-094252. PMID 40132832